CLINICAL TRIAL: NCT00169936
Title: Evaluation of Magnetocardiography as a Tool for Non-invasive Detection of Tissue Rejection in Cardiac Transplant Recipients
Brief Title: Magnetocardiography as a Non-Invasive Tool for Detecting Tissue Rejection in Heart Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CardioMag Imaging (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 20-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Heart Transplantation

INTERVENTIONS:
Device: Magnetocardiograph

SUMMARY:
Heart transplantation is a great procedure for selected patients with end-stage heart failure, but graft rejection remains a major factor limiting long-term survival despite continued advancement in the scientific skill of immunosuppression. The only reliable method used today to detect rejection is doing repeated biopsy of the heart. This is expensive, invasive, inconvenient to the patient, and associated with a significant risk of serious complications, as a piece directly from the inner surface of the patients heart is needed. The magnetocardiograph (MCG) device is an invention that may provide new means to assess changes in the heart tissue, as it may detect small changes that happen in the heart cells when they are undergoing rejection.

DETAILED DESCRIPTION:
Heart transplantation is an advantageous procedure for selected patients with end-stage heart failure. Graft rejection remains a major factor limiting long-term survival despite continued advancement in the scientific skill of immunosuppression. Hyperacute rejection occurs rarely since screening of recipient for anti-donor antibodies was introduced. Focal or diffuse acute cellular rejection is diagnosed by endomyocardial biopsy (EMB). Coronary angiography (CA) is used to monitor for allograft arteriopathy, also described as chronic rejection. Repeated endomyocardial biopsy (EMB) remains the only surveillance method available. Endomyocardial biopsy is expensive, invasive, inconvenient to the patient, and associated with a significant incidence of serious complications. The MCG device is an invention that may provide a sensitive and objective means to assess alterations in the heart tissue. Because the acute inflammatory process of rejection deleteriously affects myocyte structure and function, we hypothesize that either or both the de- and re-polarization changes will occur in the cardiac cycle with subsequent changes in the cardiac magnetic fields and may give altered readings in the affected patient over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult heart transplant recipients referred for surveillance biopsies
* Age greater than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Determine the magnetocardiographic changes in de- and/or re-polarization patterns in patients with tissue rejection relative to initial MCG reading obtained during no rejection.

SECONDARY OUTCOMES:
Determine the reproducibility of the MCG between two different recordings performed at times when rejection is histologically absent (grade 0-endomyocardial biopsy).
Differentiate the MCG results between time of grade 0 biopsy and that of the different rejection grades.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Smars, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States